CLINICAL TRIAL: NCT02899663
Title: Detection of Microbleeds With MRI (SWI Sequences) in Glioma Patients
Brief Title: MRI Detection of Microbleeds in Glioma Patients
Acronym: SWIGLI
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: NI_ALR_2016_1
Record Dates: First submitted 2016-09-09; First posted 2016-09-14 (Estimated); Last update posted 2016-09-14 (Estimated); Status verified 2016-09

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

SUMMARY:
Systematic retrospective medical chart and medical imaging file review of all patients receiving brain MRI for the follow-up of glioblastoma.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* Diagnosed with brain glioblastoma
* Receiving treatment with cranial radiotherapy and/or chemotherapy
* Having at least one follow-up MRI conducted that used a susceptibility weighted imaging sequence

Exclusion Criteria:

* Underage
* Absence of formal diagnosis of glioblastoma
* No available medical imaging file with MRI susceptibility weighted imaging sequence

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients suffering from brain glioblastoma
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2015-01; Primary Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Number of microbleeds diagnosed with MRI (susceptibility weighted imaging sequence) | At the time of each MRI conducted within 5 years after diagnosis